CLINICAL TRIAL: NCT01515722
Title: Interventions to Enhance Medication Persistence and Compliance in Patients With Overactive Bladder : 6-month, Randomized, Open-label, Multi-center Trial
Brief Title: Interventions to Enhance Medication Persistence and Compliance in Patients With Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-05-106
Record Dates: First submitted 2011-07-22; First posted 2012-01-24 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2012-01

CONDITIONS: Overactive Bladder
Keywords: Medication Persistence; Compliance; Health Education Intervention (HEI)
MeSH Terms: conditions — Urinary Bladder, Overactive; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health education intervention (HEI) (Experimental)
  Interventions: Behavioral: Health education intervention (HEI)
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Health education intervention (HEI) — * <Part 1> Understanding OAB
  * <Part 2> Behavioral/lifestyle modification
  * <Part 3> Bladder training
  * <Part 4> Understanding antimuscarinics
  Arms: Health education intervention (HEI)

SUMMARY:
Study Objectives: To explore the effectiveness of adjunctive intervention to enhance the medication compliance and persistence in patients with Overactive Bladder (OAB), thereby to improve treatment outcomes

Study Hypothesis: Health Education Intervention (HEI) can enhance the medication compliance and persistence, thereby can improve the treatment outcomes in conjunction with pharmacological therapy in OAB patients

Study Design: 6-month, randomized, open-label, multi-center trial at 13 university hospitals

DETAILED DESCRIPTION:
Treatment - Fesoterodine (Toviaz) 4 or 8mg

Interventions (2 arms)

- Arm 1: No intervention

Patients in this arm will not be given HEI in conjunction with pharmacotherapy (Toviaz) which was developed for this trial.

- Arm 2: Health education intervention (HEI)

HEI will be performed by trained study coordinators with the leaflet designed for this trial composed of 4 parts.

1. Part 1: Understanding OAB Physiology of bladder Definition, symptom and prevalence of OAB OAB in a treatable condition. There are many options that may help your symptoms. Lifestyle change Medications Bladder training Pelvic floor muscle exercise
2. Part 2: Behavioral/lifestyle modification Modification of dietary habits Limit bladder irritants- caffeine (coffee, tea, coke...), juice, chemical flavors, spicy food. etc. Altering fluid intake Weight management Learn how weight can affect their condition Stop smoking Constipation management
3. Part 3: Bladder training Timed voiding- Goal is urinating every 3 or 4 hours during the day without fear of wetting accidents.

   Urgency suppression Pelvic muscle contraction, count backwards from 100 by 7seconds, etc Pelvic floor muscle exercise Contraction (fast and slow) and relax the muscle for a count of 3. Repeat the fast and slow contractions 10 - 15 times. Do those at least 3 times a day.
4. Part 4: Understanding antimuscarinics How the medicine works How to take it Tips that may help manage side effects- dry mouth, constipation Therapy expectations
5. HEI include 3-day voiding diary for self tracking method.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18 years with OAB symptoms for ≥ 3 months
* The sum score of the OABSS ≥ 3 with the score of the question no.3 (urgency) ≥ 2
* The sum score of the OAB V8 ≥ 8

Exclusion Criteria:

* Any condition that would contraindication of anticholinergic treatment
* Symptomatic acute UTI during the run-in period
* Diagnosed or suspected interstitial cystitis
* Treatment with anticholinergic drugs within 12 months prior to Screening and persist over 3 months
* Treatment within the 14 days preceding Screening, or expected to initiate treatment during the study with any other treatment for overactive bladder.
* An indwelling catheter or practicing intermittent self-catheterization
* Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Difference in the % of patients maintaining persistence between no intervention and HEI group | 6 months
  Definition of "Maintaining Persistence"= a gap of ≤ 30 days between successive prescription fills

SECONDARY OUTCOMES:
Difference in the % of patients maintaining persistence between no intervention and HEI group | 1, 2 and 4 months
Difference in the % of the patients with the compliance rate ≥ 80% between no intervention and HEI group | 1, 2, 4, and 6 months
  Calculation of Compliance (%)= (total no. of drug prescribed - no. of remained drug)/total no. of drug prescribed x 100
Difference in the compliance rate between no intervention and HEI group | 1, 2, 4 and 6 months
Difference in changes in OAB symptoms between no intervention and HEI group | 1, 2, 4, and 6 months
  OABSS OAB-q short form questionnaire
Difference in the treatment satisfaction between no intervention and HEI group | 1, 2, 4, and 6 months
Reasons for non-persistence | 1, 2, 4, and 6 months
  Definition of non-persistence = a gap of > 30 days between successive prescription fills
  Examples
  1. Insufficient clinical response
  2. Adverse event
  3. Satisfied with treatment response
  4. Laboratory abnormality
  5. Subject died
  6. Protocol violation
  7. Lost to F/U
  8. Subject no longer willing to participate in study
  9. Pregnancy
  10. High patient out-pocket cost
  11. Others (provide detailed reason)
Adverse events | 1, 2, 4, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (13):
- South Korea (13):
  - Bucheon St. Mary's Hospital, The Catholic University of Korea, Bucheon-si
  - Bucheon Hospital, Soonchunhyang University College of Medicine, Bucheon-si
  - Samsung Changwon Hospital, Sungkyunkwan University School of Medicine, Changwon
  - Daegu Catholic University College of Medicine, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Medical School, Gwangju
  - Pusan National University Hospital, Pusan
  - Cheil General Hospital & Women's Healthcare Center, College of Medicine, Kwandong University, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Anam Hospital, College of Medicine, Korea University, Seoul
  - Asan Medical Center, Ulsan University College of Medicine, Seoul

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598